CLINICAL TRIAL: NCT06433986
Title: Management of Isolated RT 3 Gingival Recession With Modified Coronally Advanced Tunnel Versus Vestibular Incision Subperiosteal Tunnel Access With Volume Stable Collagen Matrix: A RCT
Brief Title: MCAT Versus VISTA With Volume Stable Collagen Matrix in RT3 Gingival Recession
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rohan Goyal Perio 24/35
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Gingival Recession
Keywords: gingival recession; esthetics; phenotype
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Coronally Advanced Tunnel (MCAT)Technique (Experimental): Scaling and root planing will be performed and after resolution of gingival inflammation, root coverage procedure will be done with Volume Stable Collagen Matrix(VCMX) using MCAT.
  Interventions: Procedure: Modified Coronally Advanced Tunnel (MCAT)Technique
- Vestibular Incision Subperiosteal Tunnel Access (VISTA)Technique (Active Comparator): Scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage procedure will be done with Volume Stable Collagen Matrix(VCMX) using VISTA.
  Interventions: Procedure: Vestibular Incision Subperiosteal Tunnel Access (VISTA)Technique

INTERVENTIONS:
Procedure: Modified Coronally Advanced Tunnel (MCAT)Technique — Scaling and root planing will be performed and after resolution of gingival inflammation, root coverage procedure will be done with Volume Stable Collagen Matrix(VCMX) using MCAT.
  Arms: Modified Coronally Advanced Tunnel (MCAT)Technique
Procedure: Vestibular Incision Subperiosteal Tunnel Access (VISTA)Technique — Scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage procedure will be done with Volume Stable Collagen Matrix(VCMX) using VISTA.
  Arms: Vestibular Incision Subperiosteal Tunnel Access (VISTA)Technique

SUMMARY:
This study aims to compare MCAT technique (supraperiosteal approach with coronal advancement of flap) with VISTA technique(subperiosteal approach with coronal advancement of flap), Further, it may be hypothesized that supraperiosteal placement of graft material (in MCAT technique) may be better due to better blood supply, and MCAT technique utilizes a microsurgical concept, including microsurgical blades and suture material, which improves wound healing and establishes a better esthetic result and results in better outcome in terms of root coverage percentage compared to VISTA. Therefore, this study aims to compare minimally invasive technique MCAT and VISTA using VCMX as a graft in RT3 gingival recession in anterior teeth.

DETAILED DESCRIPTION:
Gingival recession is the migration of the gingiva to a point apical to the cement-enamel junction and is considered one of the most common periodontal problems.Besides aesthetic complaints, GR may also cause root hypersensitivity, risk for development of caries or non-carious cervical lesions, and difficulties to achieve optimal plaque control. In modified coronally advanced Tunnel (MCAT) technique partial-thickness flap is created on the entire buccal aspect, no parts of the alveolar bone are exposed, and resorption of bony structures, which occurs when using a full-thickness flap can be avoided, also,it minimizes trauma and ensure a better blood supply for the graft.

Zadeh H. in 2011 introduced a conservative modification in tunnel technique; vestibular incision subperiosteal tunnel access (VISTA) which preserve the papillary integrity and enhances patients compliance. Vista technique allows gingival tissue regeneration through subperiosteal undermining of soft tissues using a vestibular incision instead of elevating the whole flap.VISTA offers broader access and maximum esthetic outcome because of placement of incision in the frenum region.

ELIGIBILITY:
INCLUSION CRITERIA-

* Patients with RT 3 isolated recession defects present Labially in Anterior teeth region,with vestibular depth>=6mm
* Systemically healthy individuals.
* Age >18 years old.
* A full mouth plaque score (FMPS) and full mouth BOP (FMBOP) < 20%
* Patient showing adequate compliance and willing to participate in the study.

EXCLUSION CRITERIA-

* Patients having systemic disease such as hypertension, diabetes, hyperthyroidism or on medication that influence the outcome of periodontal therapy.
* Previous surgical attempt to correct gingival recession.
* Crowding of affected teeth and tooth without adjacent contact teeth.
* Patients with active periodontal disease.
* Smokers and tobacco users.
* Pregnant and lactating women.
* Involved tooth with trauma from occlusion
* Involved tooth with prosthesis.
* Endodontically treated tooth.
* Tooth with cervical abrasion/undetectable CEJ/ caries.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Root coverage percentage | 6 months
  percentage of root coverage will be calculated by using pre and post operative recession depth

CONTACTS AND LOCATIONS:
Overall Officials: ROHAN GOYAL, BDS, Principal Investigator — PGIDS, Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No